CLINICAL TRIAL: NCT05264753
Title: A Multicenter, International, Prospective, Retrospective, Post Marketing Clinical Follow Up Study to Evaluate the Efficacy and Safety of the Occlutech Patent Ductus Arteriosus Occluder (PDA Occluder) in Patients With Patent Ductus Arteriosus Defects
Brief Title: Post Marketing Clinical Follow Up Study to Evaluate Efficacy and Safety of the Occlutech PDA Occluder in Patients With Patent Ductus Arteriosus Defects
Status: Recruiting | Type: Observational
Sponsor: Occlutech International AB (Industry)
Responsible Party: Sponsor
Other Study IDs: Occ2020_03
Record Dates: First submitted 2021-12-13; First posted 2022-03-03 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Patent Ductus Arteriosus
Keywords: Occlutech PDA Occluder; Patent ductus arteriosus closure; Transcatheter PDA occlusion; Percutaneous catheter-based intervention; Occluder device; Post-marketing clinical follow-up; PMCF; Prospective and retrospective study; Multicenter international study; Efficacy and safety; Echocardiography follow-up; Pediatric cardiology
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Occlutech® PDA Occluder — Non-surgical occlusion of Patent Ductus Arteriosus (PDA).

SUMMARY:
This retrospective and prospective, multicenter, international post marketing follow up study evaluates the safety and efficacy of the Occlutech® PDA Occluder, delivered using the Occlutech Occlusions Pusher (OOP), in subjects with patent ductus arteriosus (PDA) defects. Safety and efficacy assessments include vital signs, electrocardiograms, and echocardiographic evaluations performed at baseline/implantation (including assessments within 36 hours post procedure), as well as at follow up visits occurring between Day 30 and Day 90, 6 months to 1 year, 1 to 2 years, and 2 to 3 years after implantation.

DETAILED DESCRIPTION:
The Occlutech® PDA Occluder is an occlusion system designed for the percutaneous, catheter based, non surgical closure of Patent Ductus Arteriosus (PDA), and is delivered using the Occlutech Occlusions Pusher (OOP) and Occlutech Delivery Set (ODS), which are recommended as compatible delivery systems. This post marketing clinical follow up study aims to evaluate the safety and efficacy of the Occlutech® PDA Occluder in subjects with PDA. The study is designed as a retrospective and prospective, multicenter, international investigation in which safety and efficacy will be assessed through vital signs, electrocardiography, and echocardiography at baseline/implantation (including assessments performed within 36 hours post procedure), followed by evaluations at Day 30 to Day 90, 6 months to 1 year, 1 to 2 years, and 2 to 3 years after implantation. A total of 217 evaluable subjects is required to estimate a proportion of ≤10% (or ≥90%) with a precision of 4% at an alpha level of 5%, corresponding to a two sided 95% confidence interval width of ≤8%. To account for an anticipated maximum drop out rate of 15%, a total of 255 subjects will be enrolled. Approximately 90% of enrolled participants are expected to be children aged 0-10 years. The primary objective of this study is to assess the safety of the Occlutech® PDA Occluder in subjects requiring transcatheter PDA closure, while the secondary objective is to evaluate the device's efficacy in achieving successful occlusion of the PDA

ELIGIBILITY:
Inclusion Criteria:

* A subject of any age will be eligible for PDA closure if he or she meets the indication and area of application as laid down in the IFU. Including subjects more than 3 kg. Thus, the Occlutech PDA Occluder is intended for the non-surgical occlusion of Patent Ductus Arteriosus (PDA) defects.
* Male or female subjects.
* Subjects or their parents/guardians understanding the nature of the study and providing their informed consent to participation.
* Subjects willing and able to attend the follow-up visits and procedures foreseen by study CIP.

Exclusion Criteria:

Contraindications as laid down in the IFU:

* Silent ductus or serious pulmonary hypertension:
* Pulmonary Vascular Resistance (PVR) > 8 Wood Units
* Presence of a known coagulation disorder
* Thrombus at the position allocated for the implantation
* A vein thrombosis in the blood vessels chosen for the introducing system
* An active infection (active endocarditis or other infections causing bacteremia) or history of endocarditis within 3 months from the procedure.
* Nitinol intolerance (nickel or titanium)
* Contrast medium intolerance
* Subjects who have a vascular system (which is used to access the defect) that is too small to admit the required sheath

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Full Analysis Set (safety): All patients intended to be treated with PDA Full Analysis Set (efficacy): All patients with implanted PDA
Sampling Method: Non-Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2029-10-25 (Estimated); Study Completion 2029-11-25 (Estimated)

PRIMARY OUTCOMES:
Safety primary endpoint | 1 year
  The primary safety endpoint is defined as the incidence of any Serious Adverse Device Effects (SADEs) including procedure-related death, procedure-related stroke, systemic embolism, severe hemolysis, device embolization, cardiac tamponade, infective endocarditis, or vascular complications requiring surgery up to 1-year post-implantation.
Efficacy primary endpoint | 2 years
  The primary efficacy endpoint is defined as successful implantation of the Occlutech® PDA Occluder with a complete closure of the PDA (defined as >90% PDA closure represented by no or small residual flow) as assessed by echocardiography post-implantation) within 2-year post- implantation follow-up.

SECONDARY OUTCOMES:
Safety secondary endpoint | 3 years
  Secondary safety endpoints will assess all minor complications such as transient hemolysis, vascular complications not requiring surgery, or all minor complications which are deemed relevant at the discretion of each investigator. Additionally, an assessment of all Serious Adverse Events (SAE) will be included in the analyses.
Efficacy secondary endpoint | 3 years
  Secondary efficacy assessments refer to the variation in the data from baseline to 3 years after the procedure in parameters such as, but not limited to, aortic blood pressure, pulse rate, LVFS, pulmonary artery pressure, and ECG records.

CONTACTS AND LOCATIONS:
Locations (15):
- CHU Sainte-Justine, Montreal, Canada
- France (2):
  - CHU de Lille - Institut Cœur-Poumon, Lille
  - Hôpital Mère Enfant, CHU de Nantes, Nantes
- Children's Hospital Ireland at Crumlin, Dublin, Ireland
- Ospedale Pediatrico Bambino Gesù, Roma, Roma, Italy
- Rawalpindi Institute of Cardiology, Rawalpindi, Rawalpindi, Pakistan
- Children´s Hospital, Karolinska University, Stockholm, Sweden
- Insel Gruppe, Bern, Switzerland
- Tunisia (2):
  - Hospital La Rabta, Tunis
  - Military Hospital, Tunis
- Turkey (Türkiye) (4):
  - Aydın Adnan Menderes University Hospital, Aydin, Efeler
  - Eskişehir Osmangazi University Hospital, Eskişehir, Eskişehir
  - Çukurova University Hospital, Adana, Sarıçam
  - Dicle University Hospital, Diyarbakır, SUR
- Royal Brompton & Harefield Hospitals, London, London, United Kingdom